CLINICAL TRIAL: NCT06281639
Title: RAPID: a Comparison Study of a Novel Ultrasound Device of Automated Congenital Heart Imaging
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PEDS-2023-32532
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- study group: Caregivers who have a child with a scheduled Pediatric congenital ultrasound (PCU) the day of recruitment
  Interventions: Device: RAPID

INTERVENTIONS:
Device: RAPID — test the clinical screening potential for congenital heart disorders using a single ECHO image taken by the RAPID device

SUMMARY:
The RAPID ultrasound is a portable imaging device that captures a one point image from the subcostal region of the heart. The device is set on the patient's chest and captures the image in <1 minute. It uses ultrasound imaging energy that is similar to commercialized devices and safe for patients of all ages and sizes. The device is a non-significant risk and therefore will not require an IDE. Images from RAPID will be taken directly before or after the standard clinical PCU. Images taken from both the RAPID device and the standard PCU will be de-identified and stored securely in BOX for review by two independent cardiologists. Image reviews will be conducted within Box.

ELIGIBILITY:
Inclusion Criteria:

* <1 years old
* Be a patient at Masonic Children's Hospital or Masonic Children's Heart Center clinic undergoing PCU

Exclusion Criteria:

* Open Chest
* On ECMO
* Deemed medically unstable by care team
* Cardiology, ICU, hospitalist or bedside nurse concerns

Max Age: 1 Year | Sex: All
Age Groups: Child
Study Population: children with a scheduled PCU the day of recruitment
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-07-21 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
RAPID imaging quality | 30minutes
  comparing the result of the data and imaging collected from the gold standard (PCU) vs the prototype device (RAPID)
  Two independent cardiologists will review each de-identified image in a large batch of standardized images consisting of random images from both RAPID and PCU. Each image will be reviewed by the cardiologists based on a specific checklist

CONTACTS AND LOCATIONS:
Overall Officials: Gwenyth Fischer, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States